CLINICAL TRIAL: NCT03466307
Title: Comparison of Clinical and Ultrasonographic Parameters of Rotator Cuff Tendinopathy Patients With and Without Nocturnal Pain
Brief Title: Ultrasonographic Parameters and Life Quality in Nocturnal Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Çiğdem Aydoğan, Medical Doctor in Physical Medicine and Rehabilitation Clinic, Suleyman Demirel University
Other Study IDs: 198
Record Dates: First submitted 2018-02-21; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Musculoskeletal Pain
Keywords: Nocturnal pain; shoulder pain; ultrasonography; resistive index; quality of life; anterior circumflex humeral artery
MeSH Terms: conditions — Musculoskeletal Pain; Shoulder Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Thirty patients with nocturnal shoulder pain
  Interventions: Device: Ultrasonography
- Group B: Thirty patients without nocturnal shoulder pain
  Interventions: Device: Ultrasonography
- Group C: Healthy controls
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Ultrasonographic examination of shoulder

SUMMARY:
This study aimed to investigate the effects of nocturnal pain on clinical and ultrasonographic parameters in patients with rotator cuff tendinopathy.

DETAILED DESCRIPTION:
Thirty patients with nocturnal pain, 30 patients without nocturnal pain, and 30 healthy subjects were included in the study. The demographic characteristics and body mass indexes of the patients were recorded. The visual analogue scale was used to determine pain severity. The American Shoulder and Elbow Surgeons Scale Assessment, Short Form-36 and Beck Depression Inventory were used to determine patients' shoulder function, general quality of life and depression levels, respectively. The peak systolic velocity and resistive index of anterior circumflex humeral artery was assessed with power doppler ultrasonography.The peak systolic velocity and resistive index of anterior circumflex humeral artery values of the affected and unaffected sides were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years diagnosed with rotator cuff tendinopathy

Exclusion Criteria:

* Severe limitation and pain in head and neck movements
* Loss of strength
* Sensation and reflexes loss in the upper extremity
* Limitation in passive shoulder movements on physical examination
* Systemic rheumatic disease
* Diabetes mellitus
* Malignant disease
* Active infection
* Intraarticular injection
* Trauma
* Dementia
* History of surgery
* Bilateral should pain
* Psychiatric discomfort
* Smoking history
* Antiinflammatory drugs or received physical therapy within the last 3 months
* Beck depression score of higher than 13.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years diagnosed with rotator cuff tendinopathy attending our physical medicine and rehabilitation outpatient clinic and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Anterior circumflex humeral artery peak systolic velocity | 1 week
  Ultrasonographic examination
Anterior circumflex humeral artery resistive index | 1 week
  Ultrasonographic examination

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Aydoğan, Principal Investigator — Suleyman Demirel University

IPD SHARING:
Plan to Share IPD: Undecided